CLINICAL TRIAL: NCT04371133
Title: The Role of Serum Adropin, Salusin-α, Netrin-1, and Nesfatin-1 in Endometrioma and Their Association With Insulin Resistance
Brief Title: Anti-inflammatory Markers in Endometrioma
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Burak Sezgin, Principal Investigator, Muğla Sıtkı Koçman University
Other Study IDs: 22/08/2019-05
Record Dates: First submitted 2020-04-25; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Endometrioma; Inflammation
Keywords: endometrioma; adropin; salusin-α; netrin-1; nesfatin-1; insulin resistance
MeSH Terms: conditions — Endometriosis; Inflammation; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum blood samples for each participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometrioma: Endometrioma (n=23)
  Interventions: Diagnostic Test: Adropin (ng/L)
- Healthy controls: Healthy controls Healthy volunteers n=25
  Interventions: Diagnostic Test: Adropin (ng/L)

INTERVENTIONS:
Diagnostic Test: Adropin (ng/L) — Thawed samples were measured on a Molecular Devices SpectraMax i3 Multi-Mode, Microplate Reader (batch number: SER 35 370-1448, made in Austria) using enzyme linked immunosorbent assay (ELISA).
  Other Names: Salusin-α (pg/mL); Netrin-1 (pg/mL); Nesfatin-1 (ng/mL)

SUMMARY:
Investigators aimed to measure the serum levels of adropin, salusin-α, netrin-1, and nesfatin-1, anti-inflammatory effects of which have been demonstrated previously, in endometriosis patients and to find out any association of them with insulin resistance.

DETAILED DESCRIPTION:
Endometriosis is defined as the presence of endometrial gland and stroma outside the endometrial cavity affecting almost 10% of the women of reproductive age. Although benign, it disrupts the quality of life of the inflicted patients through symptoms such as dysmenorrhae, dyspareunia, chronic pelvic pain, and infertility. The pathogenesis of endometriosis has not yet been clearly elucidated, however, recent papers implies an underpinning role of inflammation There is a limited number of studies about the levels of these parameters in endometriosis and to date, no report is available on the levels of adropin and netrin-1 in endometriosis. Likewise, according to the investigator's literature search, no research explaining the association of endometriosis with insulin resistance has yet been published. In present study, in an attempt to describe inflammatory pathways playing a role in endometriosis pathogenesis, Investigators aimed to measure the levels of serum adropin, salusin-α, netrin-1, and nesfatin-1, anti-inflammatory effects of which have been priorly demonstrated, and to find out any association of them with insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

·Histopathologically confirmed diagnosis of endometrioma

Exclusion Criteria:

* Any patients with DM,
* chronic kidney disease (CKD),
* CAD,
* heart failure (HF),
* cerebrovascular accident (CVA),
* malignancy,
* rheumatoid disorder,
* liver disease, and
* active infections were excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — patients with endometrioma
Study Population: Laporoscopically and histopathologically diagnosed 23 endometrioma patients and 25 healthy individuals with no endometrioma constituting the control group were included to this study.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Serum Adropin level | preoperative in the morning or Day 1 in outpatient clinic,preprandial for healthy volunteers
  Serum Adropin level in ng/L
Salusin-α | preoperative in the morning or Day 1 in outpatient clinic, preprandial for healthy volunteers
  Serum Salusin-α level in pg/mL
Netrin-1 | preoperative in the morning or Day 1 in outpatient clinic, preprandial for healthy volunteers
  Serum Netrin-1 level in pg/mL
Nesfatin-1 | preoperative in the morning or Day 1 in outpatient clinic, preprandial for healthy volunteers
  Serum Nesfatin-1 level in ng/L

CONTACTS AND LOCATIONS:
Overall Officials: Burak Sezgin, Dr, Principal Investigator — Mugla Sıtkı Kocman University Faculty of Medicine
Locations (1):
- Mugla Sıtkı Kocman University Faculty of Medicine, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided